CLINICAL TRIAL: NCT06310577
Title: Evaluation of Leak-free Bronchoscope Adapter to Limit Ventilated Air Volume Loss and Aerosolization From Intubated Patients Who Undergo Bronchoscopy
Brief Title: Evaluation of Leak-Free Bronchoscope Adapter to Limit Ventilated Air Volume Loss During Bronchoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Katherine Su, Clinical Assistant Professor, Attending Surgeon, Endeavor Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EH23-343
Record Dates: First submitted 2024-02-19; First posted 2024-03-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Disease
Keywords: Bronchoscope adapter
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Self-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Leak free bronchoscope adapter (Experimental): As a standard part of procedure, bronchoscopy will be performed using the "standard commercial adapter". Following the standard bronchoscope adapter use, leak-free bronchoscope adapter will be tested to compare the amount, and quality of air leaked between the"standard commercial adapter" and the "leak-free adapter.
  Interventions: Device: Leak-free bronchoscope adapter

INTERVENTIONS:
Device: Leak-free bronchoscope adapter — Bronchoscopy using both a standard adapter and a leak-free adapter will be performed.

SUMMARY:
The purpose of this research is to evaluate the ability of a new bronchoscope adapter called "leak-free adapter" to limit the amount of air leaking out to the operating room (OR) from the ventilator in intubated patients who undergo bronchoscopy.

DETAILED DESCRIPTION:
Bronchoscopy is a commonly performed procedure where a camera tipped device is used to look into a patient's lung. To perform bronchoscopy, a "standard commercial adapter" is connected to the ventilator tubing, which lets the doctors use the bronchoscope.The design of the "standard commercial adapter" can cause about 20% of air to escape from the ventilator to the OR. This leaked air causes two issues: first, this can lead to lower oxygen levels and can limit the amount of time your physician can perform bronchoscopy. Second, the leaked air can lead to the spread of harmful particles like anesthesia gas to the OR. These particles can harm the staff in the operating room or spread to other patients in the hospital.

This study will compare the benefit of the "standard commercial adapter" to the newly developed "leak-free adapter". The investigational procedure being studied here is repeating the bronchoscopy with the leak-free adapter. Outcomes (which measure the benefit of the new adapter) will be measured for each adapter independently. Bronchoscopy using both devices will be performed by the physician performing the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who will be undergoing elective intubation for either a surgical or bronchoscopic procedure (diagnostic or therapeutic)
2. Both males and females
3. Adults 18 years and older

Exclusion Criteria:

1. Significant protocol deviation
2. Significant non-compliance with protocol or study requirements
3. An adverse event which requires discontinuation which results in the inability to continue to comply with study procedures.
4. Consent is withdrawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-17 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants able to undergo bronchoscopic evaluation using the "leak-free adapter" | During the bronchoscopy procedure
  Assessment of the capacity to complete the full bronchoscopic procedure using the "leak-free adapter" device.
Heart rate (bpm) | Immediately before the procedure and during the procedure
  Prior to the initiation of the bronchoscopic procedure, the patient's will heart rate will be recorded. These values will be continuously monitored and recorded throughout the bronchoscopic procedure.
Blood pressure (mmHg) | Immediately before the procedure and during the procedure
  Prior to the initiation of the bronchoscopic procedure, the patient's blood pressure will be recorded. These values will be continuously monitored and recorded throughout the bronchoscopic procedure.
Oxygenation as measured by SpO2 | Immediately before the procedure and during the procedure
  Quantification and comparison of patient oxygenation using the "leak-free bronchoscope adapter" vs. the "standard commercial adapter". A pulse oximeter will be used to measure the patient's oxygen saturation (SpO2). Prior to bronchoscopy, the patients circulating oxygen saturation will be recorded during 10 ventilated breaths. Upon initiation of bronchoscopy, the SpO2 level will be measured throughout the procedure.
Assessment of adverse events | During the procedure and immediately after the procedure
  Any adverse events related to the leak-free adapter use will be evaluated.

SECONDARY OUTCOMES:
Evaluation of bronchoscope adapter tidal volume loss efficacy | During the bronchoscopy procedure
  Quantification and comparison of the proportion of tidal volume delivered to a patient by the ventilator during bronchoscopy using the "leak-free bronchoscope adapter" vs. the "standard commercial adapter".
Evaluation of bronchoscope adapter aerosolization efficacy | During the bronchoscopy procedure
  Quantification and comparison of aerosolized gas delivered to the ambient environment by the ventilator during bronchoscopy using the "leak-free bronchoscope adapter" vs. the "standard commercial adapter".
Peak airway pressure (cmH2O) | During the bronchoscopy procedure
  Quantification and comparison of pulmonary pressure parameters by the ventilator during bronchoscopy. Peak airway pressure (cmH2O) will be obtained from ventilator during bronchoscopy using the "leak-free bronchoscope adapter" vs. the "standard commercial adapter".
Dynamic compliance (mL/CmH2O) | During the bronchoscopy procedure
  Quantification and comparison of pulmonary pressure parameters by the ventilator during bronchoscopy. Dynamic compliance (mL/CmH2O) will be obtained from ventilator during bronchoscopy using the "leak-free bronchoscope adapter" vs. the "standard commercial adapter".

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Su, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Chicago, Illinois, United States